CLINICAL TRIAL: NCT07230223
Title: Safety and Efficacy of Ev.FV in Epidermolysis Bullosa Patients, A Randomized Clinical Trial, Phase 1 , 2
Brief Title: Effect of Ev.FV on Wound Healing in Dystrophic Epidermolysis Bullosa
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Leila Dehghani, Dr. Leila Dehghani, Isfahan University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: shahid beheshti UMS
Record Dates: First submitted 2024-06-28; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Dystrophic Epidermolysis Bullosa; Wound Heal
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Qualified patients who have confirmed chronic wounds (10-50cm2) are included in the study after completing the consent form
  Interventions: Biological: Ev.FV 1.0 x 1011 par/ml

INTERVENTIONS:
Biological: Ev.FV 1.0 x 1011 par/ml — Ev.FV 1.0 x 1011 par/ml, IV, Total of 6 doses every 2weeks

SUMMARY:
Epidermolysis bullosa (EB) is a hereditary disease of skin tissues that causes painful bleeding blisters in the skin and mucous membrane. The prevalence of this disease is 1 in 50,000. The severity of the disease varies depending on the type of disease and may even lead to death. This disease is caused by a genetic mutation in keratin or collagen, and its incidence is the same in all men and women of different human races. In these patients, the skin becomes extremely fragile and peels off with the slightest scratch. Many blisters are one of the most obvious symptoms of this disease. The possibility of skin cancer in people suffering from this disease is more than others.

Nowadays, the preference of cell therapy methods is to use biological products produced by cells such as extracellular vesicles and mitochondria instead of stem cells. The use of Extracellular vesicles and engineered EVs as messenger carriers can introduce a new treatment method based on cell products for skin regeneration and as an alternative to cell therapy.

Therefore, in this study, EV.FV will be applied topically to patients.

DETAILED DESCRIPTION:
Mesenchymal stem cell-derived EV which included Five Factors act as cell-free nanovesicles that mediate intercellular communication by transferring functional biomolecules including mRNA, microRNA, proteins, and lipids to recipient skin cells. In dystrophic epidermolysis bullosa, these exosomes facilitate wound repair and regeneration through several mechanisms: (1) modulation of inflammation by down-regulating pro-inflammatory cytokines; (2) stimulation of fibroblast and keratinocyte proliferation and migration; (3) promotion of angiogenesis via vascular endothelial growth factor (VEGF) signaling; and (4) potential delivery of collagen VII related proteins and mRNAs that support dermal epidermal junction repair. Thus, the therapeutic benefit of exosome therapy arises from paracrine signaling and molecular cargo transfer rather than cell engraftment, providing a safer and more controlled alternative to live stem cell transplantation.

Our study focused on dystrophic EB (DEB), the most severe form, where loss of collagen VII disrupts anchoring fibrils and dermal-epidermal adhesion. This pathology makes DEB an appropriate target for regenerative therapies such as mesenchymal stem cell-derived EVs and investigates if EVs from MSCs are safe and effective for treating DEB. It will examine how well these exosomes help heal wounds and promote tissue regeneration, hoping to find a new biological treatment option for this challenging disease.

ELIGIBILITY:
Inclusion Criteria:

* DEB participants determined by electron microscopy, or genetic testing. Individuals with severe DEB (eg, RDEB patients with an absence of collagen VII) and milder forms of DEB (eg, RDEB patients with reduced levels of collagen VII) will be eligible.
* People with one or more active wounds (each between 10 and 50 square centimeters on the arms, legs or trunk.)
* Participants must be willing to comply with the requirements of the protocol and have consent to participate in the project.
* Participants must be negative in the urine drug screening visit.

Exclusion Criteria:

* Participants with clinical evidence of systemic infection.
* Participants have a history of bone marrow transplantation.
* Participants must have evidence of autoimmune disease, including insulin-dependent diabetes.
* Participant has evidence of significant wound healing prior to treatment (ie, wound closure ≥ 20% during treatment at the first observation period).
* Participant has a severe medical condition, such as malignancy (including skin cancer), life expectancy less than 2 years, which limits movement to the clinical center.
* Participants have a current history of alcohol or substance abuse or a history of alcohol or substance abuse that requires treatment in the past 12 months.
* People participating in the screening should have a positive hepatitis and human immunodeficiency virus (HIV) test result.
* Women who are pregnant, lactating or planning to become pregnant during the study
* Women who are of reproductive age and use birth control pills.

Ages: 3 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
Rate of wound closure | Day 14
  percentage reduction in wound area compared to baseline, assessed by digital planimetry
EBDASI | Day 14, 28, month 3 and month 6
  EBDASI: epidermolysis bullosa disease activity and scarring index; measured in percentage change to baseline score,

SECONDARY OUTCOMES:
pain score (VAS Scale) | 30 days
  Change in pain intensity at the wound site measured using VAS Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Masoud Soleimani, Prof, Study Director — Shahid Beheshti University of Medical Sciences
Locations (1):
- Alzahra Hospital, Isfahan, Iran